CLINICAL TRIAL: NCT05520827
Title: A Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Single Rising Doses of BI 1584862 Administered as Tablet to Healthy Male Subjects (SRD Part), and a Randomised, Open-label, Single-dose, Two-way Crossover Part Investigating Relative Bioavailability of BI 1584862 as Tablet With and Without Food in Healthy Male Subjects (FE Part)
Brief Title: A Study in Healthy Men to Test How Different Doses of BI 1584862 Are Tolerated and How BI 1584862 is Taken up in the Body With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1484-0001; 2022-001019-15 (EudraCT Number)
Record Dates: First submitted 2022-08-29; First posted 2022-08-30 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: SRD-Part: parallel-group design FE-Part: two-way crossover design
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Rising Dose part: BI 1584862 (Experimental)
  Interventions: Drug: BI 1584862
- Single Rising Dose part: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Food effect part: BI 1584862 fed (treatment test, T)/ BI 1584862 fasted (treatment reference, R) (Experimental)
  Interventions: Drug: BI 1584862
- Food effect part: BI 1584862 fasted (treatment reference, R)/ BI 1584862 fed (treatment test, T) (Experimental)
  Interventions: Drug: BI 1584862

INTERVENTIONS:
Drug: BI 1584862 — BI 1584862
  Arms: Food effect part: BI 1584862 fasted (treatment reference, R)/ BI 1584862 fed (treatment test, T); Food effect part: BI 1584862 fed (treatment test, T)/ BI 1584862 fasted (treatment reference, R); Single Rising Dose part: BI 1584862
Drug: Placebo — Placebo
  Arms: Single Rising Dose part: Placebo

SUMMARY:
Single Rising Dose (SRD) part:

The main objectives of the SRD part of this trial are to investigate safety, tolerability, and pharmacokinetics (PK) of BI 1584862 in healthy male subjects following oral administration of single rising doses.

Food Effect (FE) part:

The main objective of the FE part is to assess the influence of food on the relative bioavailability of the BI 1584862 tablet.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 45 years (inclusive).
* Body mass index (BMI)of 18.5 to 29.9 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular liver enzymes (AST/ALT) above upper limit of normal and creatinine exceeding 1.2 mg/dl as confirmed by repeat measurements.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair).
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension, fainting spells, or blackouts. Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
SRD-part:Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | Up to 14 days
FE-part: Area under the concentration-time curve of BI 1584862 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 6 days
FE-part: Maximum measured concentration of BI 1584862 in plasma (Cmax) | Up to 6 days

SECONDARY OUTCOMES:
SRD-Part: Area under the concentration-time curve of BI 1584862 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 6 days
SRD-Part: Maximum measured concentration of BI 1584862 in plasma (Cmax) | Up to 6 days
FE-Part: Area under the concentration-time curve of BI 1584862 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 6 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com